CLINICAL TRIAL: NCT02823873
Title: Validation of Pulsewave Oscillometric Wrist Cuff Blood Pressure Monitor in Hypertensive and Normotensive Pregnant and Postpartum Women
Brief Title: Validation of Pulsewave Blood Pressure Monitor in Hypertensive and Normotensive Pregnant and Postpartum Women
Status: Withdrawn | Type: Observational
Why Stopped: Study submitted in error
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 205588
Record Dates: First submitted 2016-06-16; First posted 2016-07-06 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension
Keywords: Hypertension; Pregnant; Preeclampsia; Gestational Hypertension; Blood Pressure; Pregnant Women; Postpartum Women
MeSH Terms: conditions — Hypertension; Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normotensive: Normotensive pregnant and postpartum women will have blood pressure measurements administered with standard clinical equipment and the Pulsewave oscillometric wrist cuff blood pressure monitor.
  Interventions: Device: Pulsewave oscillometric wrist cuff blood pressure monitor
- Hypertensive: Hypertensive pregnant and postpartum women will have blood pressure measurements administered with standard clinical equipment and the Pulsewave oscillometric wrist cuff blood pressure monitor.
  Interventions: Device: Pulsewave oscillometric wrist cuff blood pressure monitor

INTERVENTIONS:
Device: Pulsewave oscillometric wrist cuff blood pressure monitor — Blood pressure monitor utilizing wrist cuff administered and measured using mobile technology.

SUMMARY:
The purpose of this study is to test the accuracy of the Pulsewave wrist blood pressure cuff in pregnant and postpartum women who have either normal blood pressure or high blood pressure.

DETAILED DESCRIPTION:
The study will include a series of nine blood pressure measurements. The measurements will alternate between a gold standard auscultatory blood pressure measurement and the Pulsewave monitor.

A trained clinician will be used for gold standard measurements using an appropriately sized cuff around the upper arm, a sphygmomanometer, and a stethoscope. Systolic blood pressure is defined by the first Korotkoff sound; diastolic blood pressure is defined by the fifth Korotkoff sound.

Measurements by the Pulsewave monitor will be performed using a proprietary oscillometric wrist cuff automated by a computer tablet and software made by CloudDx Inc.

Women will be seated for 5 to 10 minutes before the first blood pressure measurement. During this time, 4 circumference measurements will be taken of the arm and wrist.

1. The armpit will be measured as proximally as possible.
2. The mid upper arm will be recorded by measuring at the halfway point between the acromion and the olecranon process.
3. The distal upper arm measurement will be taken approximately 2 cm proximal to the antecubital crease.
4. The wrist will be measured approximately 2 cm proximal to the wrist flexion crease.

The first two blood pressure measurements will be used as a way to orient the subject to each device and the methods so that they are comfortable with the cuff and the process. The seven subsequent measurements will be used for analysis. There will be a 30 second to 60 second period between blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or admitted to the postpartum unit
* Normotensive women - No diagnosis of hypertension
* Hypertensive women - Diagnosis of hypertensive disorder of pregnancy

Exclusion Criteria:

* Women in active labor
* Women < 18 years of age
* Non-english speakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant or postpartum women recruited from the antepartum, labor & delivery, and postpartum units of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of measurements by Pulsewave cuff that are within 5 mmHg of standard clinical measurements | Immediately after blood pressure measurement
  Test measurement will be compared to standard measurements made at the same time.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Mhyre, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be de-identified. Data may be relevant to future studies regarding mobile health technology.